CLINICAL TRIAL: NCT04503434
Title: Patients' Experiences in a Medicalized Hotel for COVID-19 Acute Care Support
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carme Hernandez, Director of Home Hospitalization unit and Coordinator of Medicalitzed-Hotel, Hospital Clinic of Barcelona
Other Study IDs: Medicalitzed Hotel COVID-19
Record Dates: First submitted 2020-06-11; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Patient Preference; COVID-19
Keywords: Hospital Hotel
MeSH Terms: conditions — Patient Preference; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 11th March 2020, the World Health Organization (WHO) declared the novel coronavirus Covid-19 as a pandemic. Urgent reorganization was required to give answers to the needs of this new illness. Since mid March, the number of patients admitted every day grew exponentially, and despite strengthening the Home Hospitalization service, resources were insufficient to care for such a number of people at home. The HH was called to transform a hotel into a medicalized healthcare space.

Current health policy emphasizes on patient experience, as one of the key components of quality of care. Analyzing patients experience will provide knowledge about their authentic concerns or what they identify as real needs, how they perceive the care received and will allow finding out if it was a good alternative. Patients must be involved in decision-making about their heath situation and treatment in order to provide an integrated healthcare.

Aims: To assess the patient experience during hospital admission in a Medicalized Hotel for COVID-19, from 8th March to 25th May, and variables that may influence these experiences.

Study type: Observational and descriptive study with a cross-sectional design. The study population consisted of patients admitted in Medicalized Hotel who met inclusion criteria.

Sample size: 517 patients. Main variable: Patient experience (collected by the Picker Patient Experience questionnaire, PPE-15, translated to Catalan and Spanish), that content four open questions analyzed in a qualitative way. Other variables: Socio-demographic and review clinical records.

DETAILED DESCRIPTION:
The current pandemic caused by the rapid spread of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) demands urgent reorganization. Hospital multidisciplinary and departmental collaboration was required to work on all the principles of overvoltage capacity, including: new space definition; provision's resources; staff recruitment; and ad hoc training. Likewise, assistant protocols suffered continuous modifications to deal with this new situation.

Catalonia is one of the 17 autonomous communities of Spain and it has been granted global competencies in the area of healthcare. The Catalan healthcare model is a multi-provider one integrated in a unique public network. The organization is structured in four integrated health areas, one of which is the Integrated Health Area of Barcelona Esquerra (Área Integral de Salud de Barcelona Esquerra - AIS-BE), caring for a population of 524,000 inhabitants, representing 35% of the population of Barcelona. The territory referred to this study, includes the Hospital Clinic as reference center, two general hospitals and 19 primary care centers. The Hospital Clínic -a tertiary university hospital- is a public institution with a long reputation of excellence in care provision, training and research at national and international level.

The management of the Hospital Clinic worked on a contingency plan, at internal and territorial level, together with the Health Department of the Generalitat de Catalunya. For the internal contingency plan to deal with the pandemic, different committees were created. Two of them were the Technical /Operational Committee and the ICU Committee. The technical committee included the Departments of Internal Medicine, Infections, Pneumology, Microbiology and all the medical and surgical departments with ICUs, occupational health, and the transversal Home Hospitalization Unit (HH) to maximize cooperation among professionals, levels of care and institutions. Hospital-at-home is defined as the service in charge of providing active treatment by health care professionals, in patient's house, for a condition that otherwise would require traditional hospitalization for a limited period of time (8). Hospital-at-home is a safe and cost effectiveness service, and has become a popular response to the increasing demand for acute hospital beds.

The idea of transforming a hotel into a healthcare facility wanted to solve three needs: a) grouping patients who required HH, b) providing more beds (offering intermediate care to patients who didn't require critical care) and c) allowing the isolation of people who cannot do it at home.

This paper consists in an observational and descriptive study with a cross-sectional design, in which we analyze patients' experience during admission in a Medicalized Hotel using a validate survey.

The study population consisted of patients admitted in Medicalized Hotel led by Hospital Clinic, Barcelona from 25th March to 8th May.

Inclusion criteria: All patients admitted in Medicalized Hospital who agreed to participate in the study Exclusion criteria: non localized or localized but rejected to participate, language barrier and dementia.

Data collection: The Picker Patient Experience Questionnaire validated into Spanish was used to measure the patient experience. The PPE-15 was developed to elicit feedback from patients to highlight aspects of care that needed improvement and to monitor performance and care.

Participants included in this analysis responded voluntarily to an online questionnaire distributed by mail, focused on their experiences around Medicalized Hotel admissions and transitional care strategies after 1 month of discharge. The questionnaire was carried out by telephone to the patients who did not have email address. The investigators, reported if the questionnaire was self-administered or by phone. The investigators used the platform "enquesta.clinic.cat" that guarantees confidentiality and security and no identification details were collected.

Other variables collected: Socio-demographic data, such as gender, age, nationality, civil status (married, single, widow/widower, in a relationship), housing status (living alone or not), educational level (compulsory school, upper secondary school or university), and employment status (still working or not), and review clinical records, like length of Medicalized Hotel stay (days of admission), inpatient's unit (those who had been in a ICU), patients discharge destination and comorbidities (Charlson Comorbidity Index). The data collected from the medical history database were encrypted and stored in an internal and safety server.

All participants were informed in advance about the aim of the study. They received all recommendations given by legal services of the Hospital Clinic and were invited to participate. The confirmation of the study participation, as well as allowing the researchers to use the information collected from medical history, will be made by clicking the link to access into the questionnaire. This study was approved by the Ethics and Investigation Committee of the Hospital Clinic (CEIm).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in Medicalized Hospital who agreed to participate in the study.

Exclusion Criteria:

* Not localized, language barrier, dementia.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 517 patients admitted to Medicalitzed Hotel with confirmed SARS-CoV2 infection from March 25th to May 8th
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
The Picker Patient Experience Questionnaire | one month
  An adapted shorter version of The Picker Patient Experience Questionnaire, validated into Spanish and Catalan was used to identify whether exist any problem in the healthcare provided. It consists of 15 questions distributed to eight dimensions of care: respect, coordination, information/communication/education, physical comfort, emotional support, involvement of relatives, transition and continuity and finally overall impression.
  The questions have from two ("yes" or "no") responses to four answer options ("yes", "yes, to some extend", "no" or "I didn't need to"). Neutral answers, such as "I did not need to", and the most positive answer are coded as a "non-problem" (score = 0). The remaining responses are coded as "problems" (score = 1). The PPE-15 has previously been found to be valid and reliable.

SECONDARY OUTCOMES:
Open questions | one month
  Four open questions were included in the questionnaire, which enclosed what worried the participants the most, which aspects did they like and which ones they dislike about the medicalized hotel and what will they improve. Those were analysed in a qualitative technique, using the MAXQDA program. This informatics program led importing, transcribing and analysing the information obtained, by keeping the most relevant data and categorising it after having done a correct codification. All the information obtained will rest anonymous.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Hernandez, PhD, Principal Investigator — Hospital Clinic
Locations (1):
- Carme Hernández, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Result] Hernandez C, Aibar J, Seijas N, Puig I, Alonso A, Garcia-Aymerich J, Roca J. Implementation of Home Hospitalization and Early Discharge as an Integrated Care Service: A Ten Years Pragmatic Assessment. Int J Integr Care. 2018 May 16;18(2):12. doi: 10.5334/ijic.3431. PMID 30127696
- [Result] Bertran MJ, Vinaras M, Salamero M, Garcia F, Graham C, McCulloch A, Escarrabill J. Spanish and Catalan translation, cultural adaptation and validation of the Picker Patient Experience Questionnaire-15. J Healthc Qual Res. 2018 Jan-Feb;33(1):10-17. doi: 10.1016/j.cali.2017.12.004. Epub 2018 Feb 14. PMID 29454739
- Available data/document: Informed Consent Form — https://enquesta.clinic.cat/index.php/admin/survey/sa/view/surveyid/818692